CLINICAL TRIAL: NCT01079182
Title: Safety and Effectiveness of Adalimumab in Patients With Ankylosing Spondylitis in Routine Clinical Practice
Brief Title: Basic Documentation of Adalimumab (Humira) in Patients With Ankylosing Spondylitis (AS)
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-147
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Daily practice; Humira; Efficacy; Safety; Ankylosing spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ankylosing spondylitis: Participants with ankylosing spondylitis

SUMMARY:
The research question explored in this study was whether the effectiveness and safety of adalimumab in participants with ankylosing spondylitis was maintained during long-term therapy in routine clinical practice in Germany.

DETAILED DESCRIPTION:
This was a postmarketing observational study (PMOS) for participants with insufficiently controlled, moderate to severe, active AS who were eligible for adalimumab therapy. Participants started treatment with adalimumab under normal clinical settings in Germany. Enrolled participants were followed during adalimumab therapy . Participants were assessed during regular clinic visits for up to 24 months and 359 clinicians (rheumatologists/orthopedists/general practitioners/internist) participated in the study. Since this was an observational trial, not all doctors followed the stated age limitations and some participants under the age of 18 were enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with active, AS for at least 4 weeks (BASDAI greater than or equal to 4).
2. Participants who failed treatment with two non-steroidal anti-inflammatory drugs (NSAIDs).
3. No contraindications for anti-tumor necrosis factors (TNF) therapy.

Exclusion Criteria:

1. Participants who do not meet the above listed inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with AS in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 4681 (Actual)
Dates: Start 2006-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Wittig, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ankylosing Spondylitis
Started | 4681
Completed | 1962
Not Completed | 2719
Not completed — Lost to Follow-up | 1634
Not completed — Adverse Drug Reaction (ADR) | 261
Not completed — Lack of Efficacy | 514
Not completed — ADR and Lack of Effectiveness | 39
Not completed — Reasons not Evaluated | 271

BASELINE CHARACTERISTICS:
Population: A total of 4681 participants enrolled in the study, but the complete set of parameters was not available for each participant (Age and gender, N=4680; duration of AS symptoms, N=4521; HLA-B27 positive, N=3807).
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 4681
Age, Continuous [Mean (Standard Deviation); unit: Years] — N= 4680 as the complete set of parameters was not available for each participant.
  Years | 43.1 (12.1)
Gender [Number; unit: Participants] — N= 4680 as the complete set of parameters was not available for each participant.
  Participants
    Female | 1620
    Male | 3060
Duration of Ankylosing Spondylitis (AS) Symptoms [Mean (Standard Deviation); unit: Years] | 14.4 (10.8)
Human Leukocyte Antigen (HLA) B27 Positive Status [Number; unit: Percentage of participants] | 84.4

OUTCOME MEASURES:

1. Secondary Outcome: Mean Number of Involved Peripheral Joints
Description: Peripheral joints were assessed by Tender Joint Counts (TJC) and Swollen Joint Counts (SJC), using pressure and joint manipulation during physical examination. Seventy-eight TJC and 76 SJC were evaluated and a score of 0 (not tender or swollen) or 1 (tender or swollen) was assigned for each joint with a higher total score indicating a greater number of involved joints.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3715
Joints
  TJC at Baseline | 3.1 (7.2)
  TJC at Month 3 (N=3576) | 1.8 (6.0)
  TJC at Month 6 (N=3172) | 1.6 (5.6)
  TJC at Month 9 (N=2821) | 1.6 (5.7)
  TJC at Month 12 (N=2583) | 1.5 (6.1)
  TJC at Month 18 (N=2162) | 1.5 (5.4)
  TJC at Month 24 (N=1804) | 1.2 (5.0)
  SJC at Baseline | 1.3 (4.5)
  SJC at Month 3 (N=3576) | 0.7 (3.4)
  SJC at Month 6 (N=3172) | 0.6 (3.0)
  SJC at Month 9 (N=2821) | 0.5 (2.9)
  SJC at Month 12 (N=2583) | 0.4 (2.3)
  SJC at Month 18 (N=2162) | 0.5 (3.1)
  SJC at Month 24 (N=1804) | 0.4 (2.3)

2. Secondary Outcome: Percentage of Participants With Extraspinal Manifestations
Description: Extraspinal manifestations (enthesitis, dactylitis, uveitis, psoriasis, and Inflammatory Bowel Disease (IBD)) were assessed by investigators and reported on the basis of their clinical evaluation and participant records.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
Percentage of participants
  Enthesitis at Baseline | 13.6
  Enthesitis at Month 3 (N=3616) | 5.6
  Enthesitis at Month 6 (N=3216) | 3.7
  Enthesitis at Month 9 (N=2858) | 4.1
  Enthesitis at Month 12 (N=2603) | 4.5
  Enthesitis at Month 18 (N=2183) | 3.5
  Enthesitis at Month 24 (N=1823) | 3.4
  Dactylitis at Baseline | 5.4
  Dactylitis at Month 3 (N=3616) | 2.4
  Dactylitis at Month 6 (N=3216) | 1.6
  Dactylitis at Month 9 (N=2858) | 1.3
  Dactylitis at Month 12 (N=2603) | 1.6
  Dactylitis at Month 18 (N=2183) | 1.3
  Dactylitis at Month 24 (N=1823) | 1.9
  Uveitis at Baseline | 3.3
  Uveitis at Month 3 (N=3616) | 1.1
  Uveitis at Month 6 (N=3216) | 0.9
  Uveitis at Month 9 (N=2858) | 0.7
  Uveitis at Month 12 (N=2603) | 0.5
  Uveitis at Month 18 (N=2183) | 0.5
  Uveitis at Month 24 (N=1823) | 0.7
  Psoriasis at Baseline | 5.4
  Psoriasis at Month 3 (N=3616) | 2.9
  Psoriasis at Month 6 (N=3216) | 2.7
  Psoriasis at Month 9 (N=2858) | 2.6
  Psoriasis at Month 12 (N=2603) | 2.5
  Psoriasis at Month 18 (N=2183) | 2.3
  Psoriasis at Month 24 (N=1823) | 2.8
  IBD at Baseline | 4.4
  IBD at Month 3 (N=3616) | 2.6
  IBD at Month 6 (N=3216) | 1.8
  IBD at Month 9 (N=2858) | 1.9
  IBD at Month 12 (N=2603) | 1.7
  IBD at Month 18 (N=2183) | 1.4
  IBD at Month 24 (N=1823) | 1.9

3. Primary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score
Description: The BASDAI was a six question, participant-reported measure of overall disease activity that probed the level of fatigue, neck/back/hip pain, peripheral joint swelling and pain, localized tenderness, as well as morning stiffness severity and duration. It was scored on a numerical rating scale that ranged from 0 (no symptoms) to 10 (severe symptoms), and the minimum clinically important difference (MCID) was 1.0. The final BASDAI score was calculated using the following equation, in which 01 - 06 represents the question number: (BASDAI01 + BASDAI02 + BASDAI03 + BASDAI04 + BASDAI05/2 + BASDAI06*1.25/2)/5. The scale for question 6 was reduced to 0-8 since BASDAI06 was multiplied by 1.25. Data are reported as the mean change total score from baseline (Month 0).
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: BASDAI score
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
BASDAI score
  Baseline | 5.5 (1.9)
  Change from Baseline at Month 3 (N=3575) | -2.0 (2.0)
  Change from Baseline at Month 6 (N=3181) | -2.1 (2.1)
  Change from Baseline at Month 9 (N=2828) | -2.2 (2.2)
  Change from Baseline at Month 12 (N=2585) | -2.3 (2.2)
  Change from Baseline at Month 18 (N=2169) | -2.3 (2.3)
  Change from Baseline at Month 24 (N=1799) | -2.3 (2.3)

4. Primary Outcome: Mean Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Score
Description: The BASFI was a ten question, participant-reported measure that evaluated physical function. Each question was scored on a numerical rating scale that ranged from 0 (no functional impairment) to 10 (maximal impairment), and the MCID was 0.7. The mean of the ten questions was the total BASFI score. Data are reported as the mean change of total score from baseline (Month 0).
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: BASFI score
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3743
BASFI score
  Baseline | 4.9 (2.4)
  Change from Baseline at Month 3 (N=3565) | -1.4 (1.9)
  Change from Baseline at Month 6 (N=3180) | -1.5 (2.0)
  Change from Baseline at Month 9 (N=2821) | -1.6 (2.1)
  Change from Baseline at Month 12 (N=2572) | -1.6 (2.1)
  Change from Baseline at Month 18 (N=2160) | -1.7 (2.2)
  Change from Baseline at Month 24 (N=1793) | -1.7 (2.2)

5. Secondary Outcome: Mean Erythrocyte Sedimentation Rate (ESR)
Description: Plasma concentrations of ESR were assessed as a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3514
mm/hour
  Baseline | 26.8 (21.6)
  At Month 3 (N=3231) | 12.9 (14.1)
  At Month 6 (N=2888) | 13.3 (15.1)
  At Month 9 (N=2540) | 13.6 (15.3)
  At Month 12 (N=2288) | 13.3 (14.1)
  At Month 18 (N=1932) | 13.3 (13.6)
  At Month 24 (N=1627) | 14.0 (13.7)

6. Secondary Outcome: Mean Plasma Concentrations of C-Reactive Protein (CRP)
Description: Plasma concentrations of CRP were assessed as a marker of systemic inflammation that provided insights into the overall anti-inflammatory effect of rheumatologic therapies.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3638
mg/L
  Baseline | 17.1 (21.8)
  At Month 3 (N=3277) | 6.2 (11.0)
  At Month 6 (N=2934) | 6.5 (13.4)
  At Month 9 (N=2601) | 6.3 (11.9)
  At Month 12 (N=2344) | 6.0 (11.9)
  At Month 18 (N=2004) | 5.5 (9.1)
  At Month 24 (N=1687) | 5.8 (9.5)

7. Secondary Outcome: Mean Bath Ankylosing Spondylitis-Global (BAS-G) Score
Description: The BAS-G was a participant-reported instrument with two items. In the first item, the participant rated the effect of their disease over the last week, and in the second item, the participant rated the effect of their disease over the previous 6 months. Each item of the BAS-G was scored on a scale ranging from 0 (no effect) to 10 (very severe effect). The mean of the two scores was the total BAS-G score and the MCID was 1.5.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: BAS-G score
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3734
BAS-G score
  Baseline | 6.7 (2.0)
  At Month 3 (N=3562) | 4.8 (2.2)
  At Month 6 (N=3178) | 4.1 (2.4)
  At Month 9 (N=2832) | 3.8 (2.4)
  At Month 12 (N=2574) | 3.6 (2.4)
  At Month 18 (N=2162) | 3.5 (2.4)
  At Month 24 (N=1796) | 3.4 (2.4)

8. Secondary Outcome: Mean Global Assessment of Disease Activity Score
Description: Global Assessment of Disease Activity was a participant-reported measure that evaluated disease activity. It was scored on a scale that ranged from 0 to 10; lower scores indicated better patient status.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3744
Score on scale
  Baseline | 6.5 (1.7)
  At Month 3 (N=3574) | 3.1 (2.1)
  At Month 6 (N=3174) | 2.8 (2.1)
  At Month 9 (N=2831) | 2.6 (2.0)
  At Month 12 (N=2574) | 2.4 (1.9)
  At Month 18 (N=2161) | 2.3 (1.9)
  At Month 24 (N=1805) | 2.2 (1.9)

9. Secondary Outcome: Mean Participant Fatigue Score
Description: Using the BASDAI questionnaire, participants assessed the overall level of fatigue/tiredness experienced by him/her. It was scored on a numerical rating scale from 0 (no symptoms) to 10 (severe symptoms).
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
Score on scale
  Baseline | 5.9 (2.3)
  At Month 3 (N=3585) | 4.3 (2.5)
  At Month 6 (N=3189) | 4.2 (2.5)
  At Month 9 (N=2837) | 4.0 (2.5)
  At Month 12 (N=2591) | 3.9 (2.5)
  At Month 18 (N=2174) | 3.8 (2.4)
  At Month 24 (N=1803) | 3.8 (2.5)

10. Secondary Outcome: Mean Participant Pain Score
Description: Using the BASDAI questionnaire, participants assessed the overall level of AS neck, back or hip pain experienced by him/her. It was scored on a numerical rating scale from 0 (no symptoms) to 10 (severe symptoms).
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
Score on scale
  Baseline | 6.7 (2.3)
  At Month 3 (N=3586) | 4.0 (2.6)
  At Month 6 (N=3191) | 3.9 (2.6)
  At Month 9 (N=2839) | 3.8 (2.6)
  At Month 12 (N=2589) | 3.7 (2.5)
  At Month 18 (N=2173) | 3.5 (2.5)
  At Month 24 (N=1804) | 3.5 (2.5)

11. Secondary Outcome: Percentage of Participants With Morning Stiffness
Description: Morning stiffness was a participant-reported assessment. The number of participants with morning stiffness were assessed at each visit.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
Percentage of participants
  Baseline | 95.4
  At Month 3 (N=3582) | 81.8
  At Month 6 (N=3186) | 79.9
  At Month 9 (N=2835) | 78.8
  At Month 12 (N=2589) | 77.6
  At Month 18 (N=2173) | 77.6
  At Month 24 (N=1802) | 77.8

12. Secondary Outcome: Mean Duration of Morning Stiffness
Description: Participants accessed the duration of morning stiffness in 15 minute intervals from 0 to 2 hours. Data are reported as the mean duration of morning stiffness ± standard deviation.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3756
minutes
  Baseline | 56.7 (34.5)
  At Month 3 (N=3582) | 33.5 (30.7)
  At Month 6 (N=3186) | 31.3 (30.0)
  At Month 9 (N=2835) | 29.6 (28.7)
  At Month 12 (N=2589) | 28.6 (28.2)
  At Month 18 (N=2173) | 27.7 (27.4)
  At Month 24 (N=1802) | 27.4 (27.0)

13. Secondary Outcome: Percentage of Participants Achieving Assessment of SpondyloArthritis International Society (ASAS) Improvement Criteria
Description: This is a four domain (participant global assessment of disease activity, assessment of spinal pain, assessment of function (BASFI), and assessment of duration/severity of morning stiffness (mean of BASDAI questions 5 and 6)), participant-reported assessment scored on a scale from 0 (best) to 10 (worst). To qualify for a 20% improvement, participants were required to have an improvement of greater than or equal to 20% and greater than or equal to 1 unit in at least 3 domains, and no worsening of greater than or equal to 20% and greater than or equal to 1 unit in the remaining domain. To achieve a 40% improvement, participants were required to have an improvement of greater than or equal to 40% and greater than or equal to 2 units in at least 3 domains, and no worsening at all in the remaining domain.
Time Frame: At 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3349
Percentage of participants
  ASAS 20 Improvement at Month 3 | 57.9
  ASAS 20 Improvement at Month 6 (N=2989) | 63.0
  ASAS 20 Improvement at Month 9 (N=2661) | 64.3
  ASAS 20 Improvement at Month 12 (N=2419) | 65.6
  ASAS 20 Improvement at Month 18 (N=2030) | 66.9
  ASAS 20 Improvement at Month 24 (N=1688) | 67.2
  ASAS 40 Improvement at Month 3 | 36.4
  ASAS 40 Improvement at Month 6 (N=2989) | 40.1
  ASAS 40 Improvement at Month 9 (N=2661) | 42.5
  ASAS 40 Improvement at Month 12 (N=2419) | 43.7
  ASAS 40 Improvement at Month 18 (N=2030) | 45.9
  ASAS 40 Improvement at Month 24 (N=1688) | 46.8

14. Primary Outcome: Number of Participants With Drug-Related Adverse Events (AEs)
Description: An adverse event/adverse experience was any reaction, side effect or other untoward event associated with the use of a drug in humans, whether or not the event was considered drug related. This included adverse events occurring from accidental or deliberate drug overdose, from drug abuse, or from drug withdrawal. Exacerbations of pre-existing conditions are also considered adverse events. Data presented are adverse events that are drug-related and are detailed in the adverse event section of this report.
Time Frame: From signing of informed consent up to 24 months
Population: Safety analysis set: Participants who received at least one dose of adalimumab.
Measure: Number; unit: Participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 4681
Participants | 1099

15. Secondary Outcome: Percentage of Participants Achieving ASAS Partial Remission Criteria
Description: This is a four domain (participant global assessment of disease activity, assessment of spinal pain, assessment of function (BASFI), and assessment of duration/severity of morning stiffness (mean of BASDAI questions 5 and 6)), participant-reported assessment scored on a scale from 0 (best) to 10 (worst). To qualify for a partial remission, participants had to have values of 2 or less (on a scale of 10) in each of the 4 domains.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3731
Percentage of participants
  Baseline | 1.1
  Month 3 (N=3537) | 17.7
  Month 6 (N=3128) | 21.5
  Month 9 (N=2785) | 23.3
  Month 12 (N=2535) | 23.9
  Month 18 (N=2132) | 24.9
  Month 24 (N=1782) | 26.8

16. Secondary Outcome: Percentage of Participants With Impairment in Daily Activities During the Last 4 Weeks
Description: The impairment of daily activities was based on participant recall of events that occurred over the 4 weeks before the visit. Percentage of participants with impairment for 0, less than 7, 7 to 14, and greater than 14 days was assessed.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3654
Percentage of participants
  0 Days at Baseline | 23.0
  0 Days at Month 3 (N=3496) | 47.2
  0 Days at Month 6 (N=3121) | 52.6
  0 Days at Month 9 (N=2793) | 55.9
  0 Days at Month 12 (N=2524) | 57.1
  0 Days at Month 18 (N=2130) | 60.2
  0 Days at Month 24 (N=1766) | 60.9
  Less Than 7 Days at Baseline | 28.5
  Less Than 7 Days at Month 3 (N=3496) | 30.3
  Less Than 7 Days at Month 6 (N=3121) | 28.5
  Less Than 7 Days at Month 9 (N=2793) | 27.2
  Less Than 7 Days at Month 12 (N=2524) | 27.2
  Less Than 7 Days at Month 18 (N=2130) | 24.4
  Less Than 7 Days at Month 24 (N=1766) | 24.0
  7 to 14 Days at Baseline | 23.4
  7 to 14 Days at Month 3 (N=3496) | 11.6
  7 to 14 Days at Month 6 (N=3121) | 9.9
  7 to 14 Days at Month 9 (N=2793) | 9.6
  7 to 14 Days at Month 12 (N=2524) | 8.9
  7 to 14 Days at Month 18 (N=2130) | 8.8
  7 to 14 Days at Month 24 (N=1766) | 8.9
  Greater Than 14 Days at Baseline | 25.1
  Greater Than 14 Days at Month 3 (N=3496) | 11.0
  Greater Than 14 Days at Month 6 (N=3121) | 9.0
  Greater Than 14 Days at Month 9 (N=2793) | 7.3
  Greater Than 14 Days at Month 12 (N=2524) | 6.8
  Greater Than 14 Days at Month 18 (N=2130) | 6.6
  Greater Than 14 Days at Month 24 (N=1766) | 6.1

17. Secondary Outcome: Percentage of Participants Who Missed Work Days Due to Ankylosing Spondylitis (AS) in the Previous 12 Months
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 2217
Percentage of participants
  Baseline | 45.7
  At Month 3 (N=2082) | 39.3
  At Month 6 (N=1870) | 32.2
  At Month 9 (N=1673) | 26.3
  At Month 12 (N=1549) | 21.3
  At Month 18 (N=1331) | 17.2
  At Month 24 (N=1105) | 14.2

18. Secondary Outcome: Mean Missed Work Days Due to Ankylosing Spondylitis in the Previous 12 Months
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 2217
Days
  Baseline | 48.0 (69.1)
  At Month 3 (N=2082) | 52.2 (74.3)
  At Month 6 (N=1870) | 56.0 (85.7)
  At Month 9 (N=1673) | 50.5 (81.7)
  At Month 12 (N=1549) | 48.0 (80.1)
  At Month 18 (N=1331) | 35.3 (61.4)
  At Month 24 (N=1105) | 35.4 (61.3)

19. Secondary Outcome: Percentage of Participants With In-Patient Hospitalization Due to Ankylosing Spondylitis in the Previous 12 Months
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3692
Percentage of participants
  Baseline | 20.6
  At Month 3 (N=3521) | 18.9
  At Month 6 (N=3134) | 16.9
  At Month 9 (N=2798) | 12.9
  At Month 12 (N=2538) | 8.4
  At Month 18 (N=2133) | 4.7
  At Month 24 (N=1762) | 3.8

20. Secondary Outcome: Mean Days of In-Patient Hospitalization Due to Ankylosing Spondylitis in the Previous 12 Months
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3692
Days
  Baseline | 16.0 (14.7)
  At Month 3 (N=3521) | 15.1 (12.6)
  At Month 6 (N=3134) | 16.3 (21.5)
  At Month 9 (N=2798) | 17.2 (26.4)
  At Month 12 (N=2538) | 18.8 (33.9)
  At Month 18 (N=2133) | 17.7 (12.4)
  At Month 24 (N=1762) | 15.3 (11.9)

21. Secondary Outcome: Percentage of Participants on Adalimumab Monotherapy
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3744
Percentage of participants
  Baseline | 78.8
  At Month 3 (N=3591) | 81.6
  At Month 6 (N=3202) | 82.8
  At Month 9 (N=2848) | 83.2
  At Month 12 (N=2598) | 83.6
  At Month 18 (N=2179) | 83.7
  At Month 24 (N=1816) | 84.6

22. Secondary Outcome: Percentage of Participants With Concomitant Non-Biologic Disease-modifying Antirheumatic Drugs (DMARDs)
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3744
Percentage of participants
  Methotrexate at Baseline | 13.0
  Methotrexate at Month 3 (N=3591) | 11.9
  Methotrexate at Month 6 (N=3202) | 11.9
  Methotrexate at Month 9 (N=2848) | 11.6
  Methotrexate at Month 12 (N=2598) | 11.5
  Methotrexate at Month 18 (N=2179) | 11.6
  Methotrexate at Month 24 (N=1816) | 11.0
  Sulfasalazine at Baseline | 7.5
  Sulfasalazine at Month 3 (N=3591) | 5.2
  Sulfasalazine at Month 6 (N=3202) | 4.2
  Sulfasalazine at Month 9 (N=2848) | 3.9
  Sulfasalazine at Month 12 (N=2598) | 3.8
  Sulfasalazine at Month 18 (N=2179) | 3.7
  Sulfasalazine at Month 24 (N=1816) | 3.3
  Other DMARDs at Baseline | 2.3
  Other DMARDs at Month 3 (N=3591) | 1.9
  Other DMARDs at Month 6 (N=3202) | 1.8
  Other DMARDs at Month 9 (N=2848) | 2.0
  Other DMARDs at Month 12 (N=2598) | 1.8
  Other DMARDs at Month 18 (N=2179) | 1.6
  Other DMARDs at Month 24 (N=1816) | 1.5

23. Secondary Outcome: Percentage of Participants With Concomitant Pain Relief/Anti-Inflammatory Agents
Description: Participants with concomitant pain relief/anti-inflammatory agents like analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase-2 (COX-2) inhibitors, and systemic glucocorticoids were assessed during the study period.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Number; unit: Percentage of participants
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3744
Percentage of participants
  Analgesics at Baseline | 17.5
  Analgesics at Month 3 (N=3591) | 12.4
  Analgesics at Month 6 (N=3202) | 11.8
  Analgesics at Month 9 (N=2848) | 11.1
  Analgesics at Month 12 (N=2598) | 11.2
  Analgesics at Month 18 (N=2179) | 10.1
  Analgesics at Month 24 (N=1816) | 10.3
  NSAIDs at Baseline | 52.3
  NSAIDs at Month 3 (N=3591) | 36.1
  NSAIDs at Month 6 (N=3202) | 33.5
  NSAIDs at Month 9 (N=2848) | 31.4
  NSAIDs at Month 12 (N=2598) | 30.2
  NSAIDs at Month 18 (N=2179) | 31.3
  NSAIDs at Month 24 (N=1816) | 30.2
  COX-2 Inhibitors at Baseline | 21.4
  COX-2 Inhibitors at Month 3 (N=3591) | 16.5
  COX-2 Inhibitors at Month 6 (N=3202) | 15.4
  COX-2 Inhibitors at Month 9 (N=2848) | 15.0
  COX-2 Inhibitors at Month 12 (N=2598) | 14.5
  COX-2 Inhibitors at Month 18 (N=2179) | 14.0
  COX-2 Inhibitors at Month 24 (N=1816) | 13.3
  Systemic Glucocorticoids at Baseline | 22.9
  Systemic Glucocorticoids at Month 3 (N=3591) | 15.2
  Systemic Glucocorticoids at Month 6 (N=3202) | 13.1
  Systemic Glucocorticoids at Month 9 (N=2848) | 11.8
  Systemic Glucocorticoids at Month 12 (N=2598) | 11.9
  Systemic Glucocorticoids at Month 18 (N=2179) | 11.3
  Systemic Glucocorticoids at Month 24 (N=1816) | 11.0

24. Secondary Outcome: Mean Equivalent Dose of Prednisolone
Description: The mean equivalent dose of prednisolone was calculated based on the International Standard for comparison of different glucocorticoid products.
Time Frame: At Baseline (Month 0), 3, 6, 9, 12, 18, and 24 months
Population: Full analysis set: Participants with adequate data available for evaluation of effectiveness.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Ankylosing Spondylitis
Number analyzed (Participants) | 3744
mg/day
  Baseline | 10.5 (15.2)
  At Month 3 (N=3591) | 6.6 (5.0)
  At Month 6 (N=3202) | 6.8 (6.6)
  At Month 9 (N=2848) | 6.4 (6.1)
  At Month 12 (N=2598) | 7.2 (14.9)
  At Month 18 (N=2179) | 6.0 (7.0)
  At Month 24 (N=1816) | 5.6 (3.8)

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 24 months
Description: Drug related AEs and all serious adverse events (SAEs) were collected during the study period.
Arm/Group | Ankylosing Spondylitis
Serious Adverse Events (participants affected / at risk) | 141/4681
Other Adverse Events (participants affected / at risk) | 1099/4681
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ankylosing Spondylitis (N=4681)
Hospitalization (Surgical and medical procedures) | 10
Hip arthroplasty (Surgical and medical procedures) | 4
Knee arthroplasty (Surgical and medical procedures) | 3
Intervertebral disc operation (Surgical and medical procedures) | 2
Surgery (Surgical and medical procedures) | 2
Vascular bypass graft (Surgical and medical procedures) | 2
Adhesiolysis (Surgical and medical procedures) | 1
Caecum operation (Surgical and medical procedures) | 1
Cardioversion (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Coronary revascularization (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Gastric operation (Surgical and medical procedures) | 1
Hernia repair (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Kidney ablation (Surgical and medical procedures) | 1
Meniscus operation (Surgical and medical procedures) | 1
Rehabilitation therapy (Surgical and medical procedures) | 1
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 1
Shoulder operation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Therapeutic procedure (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Pneumonia (Infections and infestations) | 5
Cellulitis (Infections and infestations) | 3
Acute tonsillitis (Infections and infestations) | 2
Tuberculosis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Fungal oesophagitis (Infections and infestations) | 1
Gastroenteritis escherichia coli (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pancreatitis bacterial (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Salmonellosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Stitch abscess (Infections and infestations) | 1
Systemic mycosis (Infections and infestations) | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Toe deformity (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pancreatitis (Gastrointestinal disorders) | 2
Tooth loss (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatic mass (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 2
Accident (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Haemothorax (Injury, poisoning and procedural complications) | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Ureteric injury (Injury, poisoning and procedural complications) | 1
Acute myocardial infarction (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Pyrexia (General disorders) | 4
Abasia (General disorders) | 1
Adhesion (General disorders) | 1
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 1
Disease recurrence (General disorders) | 1
Pain (General disorders) | 1
Performance status decreased (General disorders) | 1
Dizziness (Nervous system disorders) | 3
Cerebrovascular accident (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 2
Altered state of consciousness (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Multiple sclerosis (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Plantar erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Body temperature increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Laparoscopy (Investigations) | 1
Weight decreased (Investigations) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 2
Mental disorder (Psychiatric disorders) | 1
Panic disorder with agoraphobia (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Cholecystitis (Hepatobiliary disorders) | 1
Hepatocellular damage (Hepatobiliary disorders) | 1
Chondrodystrophy (Congenital, familial and genetic disorders) | 1
Factor V deficiency (Congenital, familial and genetic disorders) | 1
Conjunctivitis (Eye disorders) | 1
Visual disturbance (Eye disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Renal colic (Renal and urinary disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Adnexa uteri cyst (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Death (General disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ankylosing Spondylitis (N=4681)
Drug ineffective (General disorders) | 210
Influenza like illness (General disorders) | 50
Pyrexia (General disorders) | 33
Injection site erythema (General disorders) | 32
Fatigue (General disorders) | 27
Injection site pruritus (General disorders) | 15
Injection site irritation (General disorders) | 12
Injection site reaction (General disorders) | 12
Oedema peripheral (General disorders) | 10
Injection site pain (General disorders) | 8
Injection site swelling (General disorders) | 8
Impaired healing (General disorders) | 7
Drug intolerance (General disorders) | 5
Malaise (General disorders) | 5
Pain (General disorders) | 5
Chills (General disorders) | 4
General physical health deterioration (General disorders) | 4
Inflammation (General disorders) | 4
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 2
Condition aggravated (General disorders) | 2
Injection site rash (General disorders) | 2
Injection site warmth (General disorders) | 2
Local swelling (General disorders) | 2
Mucosal dryness (General disorders) | 2
Sensation of foreign body (General disorders) | 2
Swelling (General disorders) | 2
Abasia (General disorders) | 1
Adverse event (General disorders) | 1
Cyst (General disorders) | 1
Feeling abnormal (General disorders) | 1
Feeling cold (General disorders) | 1
Feeling hot (General disorders) | 1
Gait disturbance (General disorders) | 1
Induration (General disorders) | 1
Injection site discharge (General disorders) | 1
Injection site induration (General disorders) | 1
Injection site inflammation (General disorders) | 1
Injection site urticaria (General disorders) | 1
Mucosal haemorrhage (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Performance status decreased (General disorders) | 1
Tenderness (General disorders) | 1
Bronchitis (Infections and infestations) | 46
Upper respiratory tract infection (Infections and infestations) | 46
Nasopharyngitis (Infections and infestations) | 37
Infection (Infections and infestations) | 36
Sinusitis (Infections and infestations) | 33
Respiratory tract infection (Infections and infestations) | 24
Herpes zoster (Infections and infestations) | 15
Gastrointestinal infection (Infections and infestations) | 12
Infection in an immunocompromised host (Infections and infestations) | 12
Rash pustular (Infections and infestations) | 11
Otitis media (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 10
Acute tonsillitis (Infections and infestations) | 9
Cystitis (Infections and infestations) | 9
Oral herpes (Infections and infestations) | 9
Rhinitis (Infections and infestations) | 6
Tonsillitis (Infections and infestations) | 6
Erysipelas (Infections and infestations) | 4
Folliculitis (Infections and infestations) | 4
Furuncle (Infections and infestations) | 4
Herpes virus infection (Infections and infestations) | 4
Laryngitis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Viral infection (Infections and infestations) | 3
Vulvovaginal mycotic infection (Infections and infestations) | 3
Abscess (Infections and infestations) | 2
Bronchopneumonia (Infections and infestations) | 2
Chronic sinusitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 2
Ear infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Paronychia (Infections and infestations) | 2
Respiratory tract infection viral (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Abdominal wall abscess (Infections and infestations) | 1
Abscess jaw (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Anogenital warts (Infections and infestations) | 1
Body tinea (Infections and infestations) | 1
Borrelia infection (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Campylobacter intestinal infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Eczema impetiginous (Infections and infestations) | 1
Erythema infectiosum (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastrointestinal fungal infection (Infections and infestations) | 1
Genital abscess (Infections and infestations) | 1
Genitourinary tract infection (Infections and infestations) | 1
Gingival infection (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Infectious mononucleosis (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Latent tuberculosis (Infections and infestations) | 1
Legionella infection (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Oropharyngitis fungal (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pseudofolliculitis barbae (Infections and infestations) | 1
Puncture site abscess (Infections and infestations) | 1
Scarlet fever (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Sialoadenitis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vaginal abscess (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 35
Psoriasis (Skin and subcutaneous tissue disorders) | 30
Pruritus (Skin and subcutaneous tissue disorders) | 26
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 19
Erythema (Skin and subcutaneous tissue disorders) | 18
Alopecia (Skin and subcutaneous tissue disorders) | 13
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 12
Urticaria (Skin and subcutaneous tissue disorders) | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8
Night sweats (Skin and subcutaneous tissue disorders) | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7
Acne (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5
Rash papular (Skin and subcutaneous tissue disorders) | 5
Skin reaction (Skin and subcutaneous tissue disorders) | 5
Drug eruption (Skin and subcutaneous tissue disorders) | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 4
Skin disorder (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 2
Neurodermatitis (Skin and subcutaneous tissue disorders) | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2
Acrodermatitis (Skin and subcutaneous tissue disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Erythema annulare (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin fibrosis (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 1
Skin warm (Skin and subcutaneous tissue disorders) | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria generalised (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 17
Periodontitis (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 5
Gastrointestinal pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 4
Tooth disorder (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain lower (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gingival bleeding (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 2
Oral discomfort (Gastrointestinal disorders) | 2
Reflux oesophagitis (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 1
Diverticulum (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastroduodenitis (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Lip blister (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oedema mouth (Gastrointestinal disorders) | 1
Oral mucosal blistering (Gastrointestinal disorders) | 1
Oral mucosal disorder (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Salivary gland disorder (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Tongue black hairy (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 37
Dizziness (Nervous system disorders) | 19
Paraesthesia (Nervous system disorders) | 10
Carpal tunnel syndrome (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 4
Disturbance in attention (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 3
Burning sensation (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 2
Multiple sclerosis (Nervous system disorders) | 2
Sensory disturbance (Nervous system disorders) | 2
Ageusia (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Aphonia (Nervous system disorders) | 1
Arachnoid cyst (Nervous system disorders) | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Cluster headache (Nervous system disorders) | 1
Dysaesthesia (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Ulnar tunnel syndrome (Nervous system disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4
Limb discomfort (Musculoskeletal and connective tissue disorders) | 3
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3
Osteitis (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2
Toe deformity (Musculoskeletal and connective tissue disorders) | 2
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1
Hospitalisation (Surgical and medical procedures) | 8
Dental operation (Surgical and medical procedures) | 5
Hip arthroplasty (Surgical and medical procedures) | 5
Antibiotic prophylaxis (Surgical and medical procedures) | 4
Hip surgery (Surgical and medical procedures) | 4
Surgery (Surgical and medical procedures) | 4
Meniscus operation (Surgical and medical procedures) | 3
Tonsillectomy (Surgical and medical procedures) | 3
Arthrodesis (Surgical and medical procedures) | 2
Dental treatment (Surgical and medical procedures) | 2
Hysterectomy (Surgical and medical procedures) | 2
Inguinal hernia repair (Surgical and medical procedures) | 2
Knee operation (Surgical and medical procedures) | 2
Nasal septal operation (Surgical and medical procedures) | 2
Tendon operation (Surgical and medical procedures) | 2
Tooth extraction (Surgical and medical procedures) | 2
Allergenic desensitisation procedure (Surgical and medical procedures) | 1
Anorectal operation (Surgical and medical procedures) | 1
Aortic valve replacement (Surgical and medical procedures) | 1
Appendicectomy (Surgical and medical procedures) | 1
Arthroscopic surgery (Surgical and medical procedures) | 1
Cervical conisation (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Chondroplasty (Surgical and medical procedures) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Dental implantation (Surgical and medical procedures) | 1
Eye laser surgery (Surgical and medical procedures) | 1
Female genital operation (Surgical and medical procedures) | 1
Haemorrhoid operation (Surgical and medical procedures) | 1
Heart valve operation (Surgical and medical procedures) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
Intestinal operation (Surgical and medical procedures) | 1
Joint irrigation (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Large intestine operation (Surgical and medical procedures) | 1
Laryngeal operation (Surgical and medical procedures) | 1
Meniscus removal (Surgical and medical procedures) | 1
Oophorectomy (Surgical and medical procedures) | 1
Otorhinolaryngological surgery (Surgical and medical procedures) | 1
Radiotherapy (Surgical and medical procedures) | 1
Salpingectomy (Surgical and medical procedures) | 1
Sigmoidectomy (Surgical and medical procedures) | 1
Sinus operation (Surgical and medical procedures) | 1
Skin operation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Testicular operation (Surgical and medical procedures) | 1
Toe operation (Surgical and medical procedures) | 1
Uterine dilation and curettage (Surgical and medical procedures) | 1
Hepatic enzyme increased (Investigations) | 16
Weight decreased (Investigations) | 11
Transaminases increased (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 8
Weight increased (Investigations) | 8
Gamma-glutamyltransferase increased (Investigations) | 4
Arthroscopy (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 3
Blood pressure increased (Investigations) | 3
C-reactive protein increased (Investigations) | 2
Antinuclear antibody increased (Investigations) | 1
Biopsy breast normal (Investigations) | 1
Blood count abnormal (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood testosterone decreased (Investigations) | 1
Blood urine present (Investigations) | 1
Borrelia burgdorferi serology positive (Investigations) | 1
Computerised tomogram thorax abnormal (Investigations) | 1
Double stranded DNA antibody (Investigations) | 1
Endoscopic retrograde cholangiopancreatography (Investigations) | 1
Haematology test (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Hysteroscopy (Investigations) | 1
Laboratory test abnormal (Investigations) | 1
Lipase increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Prothrombin time shortened (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1
Visual disturbance (Eye disorders) | 10
Iritis (Eye disorders) | 7
Eye pain (Eye disorders) | 4
Dry eye (Eye disorders) | 3
Uveitis (Eye disorders) | 3
Conjunctivitis (Eye disorders) | 2
Eye inflammation (Eye disorders) | 2
Eye pruritus (Eye disorders) | 2
Iridocyclitis (Eye disorders) | 2
Ocular hyperaemia (Eye disorders) | 2
Blepharospasm (Eye disorders) | 1
Cataract (Eye disorders) | 1
Chalazion (Eye disorders) | 1
Conjunctival hyperaemia (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Myopia (Eye disorders) | 1
Ocular discomfort (Eye disorders) | 1
Sicca syndrome (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Depression (Psychiatric disorders) | 8
Depressed mood (Psychiatric disorders) | 7
Sleep disorder (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 3
Loss of libido (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 2
Emotional distress (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 2
Somatisation disorder (Psychiatric disorders) | 2
Binge eating (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Mental disorder (Psychiatric disorders) | 1
Nervousness (Psychiatric disorders) | 1
Panic disorder (Psychiatric disorders) | 1
Psychosomatic disease (Psychiatric disorders) | 1
Somatoform disorder (Psychiatric disorders) | 1
Accident (Injury, poisoning and procedural complications) | 3
Tendon rupture (Injury, poisoning and procedural complications) | 3
Accident at work (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Limb traumatic amputation (Injury, poisoning and procedural complications) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 2
Muscle injury (Injury, poisoning and procedural complications) | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Open fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Arrhythmia (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 3
Pericarditis (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 2
Cardiovascular disorder (Cardiac disorders) | 2
Coronary artery disease (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Aortic valve incompetence (Cardiac disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 21
Haematoma (Vascular disorders) | 4
Hypertension (Vascular disorders) | 4
Thrombosis (Vascular disorders) | 4
Lymphoedema (Vascular disorders) | 3
Hot flush (Vascular disorders) | 2
Blood pressure fluctuation (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Temporal arteritis (Vascular disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 6
Menorrhagia (Reproductive system and breast disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 2
Breast cyst (Reproductive system and breast disorders) | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1
Hypomenorrhoea (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Orchitis noninfective (Reproductive system and breast disorders) | 1
Prostatic disorder (Reproductive system and breast disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Anaemia neonatal (Blood and lymphatic system disorders) | 1
Haemolysis (Blood and lymphatic system disorders) | 1
Haemolysis neonatal (Blood and lymphatic system disorders) | 1
Lymphatic disorder (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Platelet disorder (Blood and lymphatic system disorders) | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Xanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 6
Anaphylactic reaction (Immune system disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Leukocyturia (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 2
Calculus ureteric (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 3
Deafness unilateral (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1
Podagra (Metabolism and nutrition disorders) | 1
Pregnancy of partner (Social circumstances) | 4
Miscarriage of partner (Social circumstances) | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.